CLINICAL TRIAL: NCT03697265
Title: A Phase II, Randomised, Double-blind, Placebo-controlled, Parallel Group, Multicentre Study Investigating Efficacy and Safety of Sepranolone (UC1010) in Patients With Premenstrual Dysphoric Disorder (PMDD)
Brief Title: A Study of Efficacy and Safety of Sepranolone (UC1010) in Patients With Premenstrual Dysphoric Disorder (PMDD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asarina Pharma (Industry)
Collaborators: Ergomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UM203
Record Dates: First submitted 2018-09-28; First posted 2018-10-05 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Premenstrual Dysphoric Disorder
MeSH Terms: conditions — Premenstrual Dysphoric Disorder | interventions — Pregnanolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sepranolone (UC1010) low dose (Experimental): Sepranolone (UC1010) low dose administered subcutaneously (SC) during the luteal phase
  Interventions: Drug: Sepranolone (UC1010) low dose
- Sepranolone (UC1010) high dose (Experimental): Sepranolone (UC1010) high dose administered subcutaneously (SC) during the luteal phase
  Interventions: Drug: Sepranolone (UC1010) high dose
- Placebo (Placebo Comparator): Placebo administered subcutaneously (SC) during the luteal phase
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sepranolone (UC1010) low dose — Subcutaneous (SC) administration
  Arms: Sepranolone (UC1010) low dose
Drug: Sepranolone (UC1010) high dose — Subcutaneous (SC) administration
  Arms: Sepranolone (UC1010) high dose
Drug: Placebo — Subcutaneous (SC) adminstration
  Arms: Placebo

SUMMARY:
The objective of this phase IIb study is to evaluate the effect and safety of Sepranolone (UC1010) on premenstrual symptoms in women with Premenstrual Dysphoric Disorder (PMDD). Patients will be taking Sepranolone or Placebo (blinded to patient and study doctor) during the two weeks preceding the menstruation of three menstrual cycles. Effect (change from baseline) will be assessed by comparison of symptoms recorded daily by the patients using a validated rating scale for assessment of PMDD symptoms. Sepranolone is an endogenous steroid.

DETAILED DESCRIPTION:
The objective of this phase IIb study is to evaluate the effect and safety of two doses of Sepranolone (UC1010) on premenstrual symptoms in women with Premenstrual Dysphoric Disorder (PMDD) in comparison to placebo, administrated during the luteal phase of three consecutive menstrual cycles. Effect will be assessed by comparison of symptoms recorded daily by the patients using a validated rating scale for assessment of PMDD symptoms and impairment of symptoms on daily life of the patients. The scale is Daily Record of Severity of Problems (DRSP). Preceding the treatment period, the diagnosis of PMDD will be established in the study participants by at lest two menstrual cycles of prospective DRSP ratings by the patients. This period will also constitute the baseline data. The effect of study medication will be assessed as the change in symptoms from baseline to during treatment. The Total symptom score of the DRSP will constitute the primary variable and the late luteal phase ratings in the respective menstrual cycles, before and during treatment, will be used.

The study will also include a follow-up (no treatment) cycle before patients final visit.

The study is conducted in four European countries (Sweden, Germany, Poland and United Kingdom) and will include up to 225 patients.

ELIGIBILITY:
Main Inclusion Criteria:

* have PMDD according to DSM-5 verified in two menstrual cycles
* have a regular menstrual cycle of 24-35 days cycle,
* use double barrier contraception, non-hormonal IUD, be truly sexually abstinent, or subject or her partner has been surgically sterilized,

Main Exclusion Criteria:

* steroid hormonal treatment or treatment with psychopharmaceuticals during previous three months
* treatments for premenstrual syndrome (PMS) or PMDD
* history of or significant medical condition ongoing
* be pregnant or plan a pregnancy within the study period

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Woman with regular menstrual cycles
Enrollment: 475 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Effect on DRSP Total symptom score | Baseline luteal phase score (average from two menstrual cycles) vs. luteal phase score during treatment.
  Change in DRSP Total symptom score (Daily Record of Severity of Problems) measured during the luteal phase (i.e. the week before menstruation) before and during treatment

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Starting from first dose given until 1 months after treatment stop
  Recording of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Shaughn O'Brien, MD, Principal Investigator — Obstetrics and Gynaecology Keele University School of Medicine and University Hospitals of North Staffordshire
Locations (12):
- Germany (5):
  - Zentrum für Klinische Forschnung, Bad Homburg
  - Emovis, Berlin
  - Medizentrum Essen Borbeck, Essen
  - Klinische Forschung Karlsruhe GmbH, Karlsruhe
  - Praxis Dr. Steinwachs, Nuremberg
- Poland (3):
  - Centrum Kliniczno-Badawcze, Elblag
  - Centrum Medyczne Angelius Provita, Katowice
  - ProCreative, Krakow
- Karolinska University Hospital, Stockholm, Sweden
- United Kingdom (3):
  - Liverpool Women's NHS Foundation Trust, Liverpool
  - Imperial College London, London
  - Obstetrics and Gynaecology Keele University School of Medicine and University Hospitals of North Staffordshire, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bixo M, Ekberg K, Poromaa IS, Hirschberg AL, Jonasson AF, Andreen L, Timby E, Wulff M, Ehrenborg A, Backstrom T. Treatment of premenstrual dysphoric disorder with the GABAA receptor modulating steroid antagonist Sepranolone (UC1010)-A randomized controlled trial. Psychoneuroendocrinology. 2017 Jun;80:46-55. doi: 10.1016/j.psyneuen.2017.02.031. Epub 2017 Mar 1. PMID 28319848